CLINICAL TRIAL: NCT06228521
Title: Efficacy and Safety of 980nm Diode Laser Versus Liquid Nitrogen Cryotherapy for the Treatment of Plantar Warts
Brief Title: Efficacy & Safety of 980nm Diode Laser vs. Cryotherapy for Plantar Warts
Acronym: LAVsCryWarts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2022-2023/080
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Warts of Foot
Keywords: cryotherapy; laser therapy; papillomaviridae; plantar warts; randomised clinical trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental): LASEmaR MINI 980 nm
  Interventions: Other: 980nm diode laser applied
- Cryotherapy group: (Active Comparator): CryoIQ
  Interventions: Other: Liquid nitrogen sprayed

INTERVENTIONS:
Other: Liquid nitrogen sprayed — Liquid nitrogen sprayed on each wart using a standardised technique. Freeze-thaw cycle repeated up to 3 times per wart per session. 4 sessions at weekly intervals.
  Arms: Cryotherapy group:
Other: 980nm diode laser applied — 980nm diode laser applied to each wart for 5 seconds at 2W power and 1mm spot size. 4 sessions at weekly intervals.
  Arms: Laser Group

SUMMARY:
The goal of this clinical trial is to compare and test the efficacy of two treatments for plantar warts. The main questions it aims to answer are:

Which treatment has a higher cure rate for eliminating plantar warts? Which treatment causes less pain during the procedure?

Participants with plantar warts will:

Be randomly assigned to receive either cryotherapy or laser therapy Undergo 4 treatment sessions at weekly intervals Have their warts assessed for complete clearance after treatment Rate their pain levels during each session

Researchers will compare the cryotherapy and laser therapy groups to see if there are differences in:

Rates of complete wart clearance Pain levels reported during treatment Adverse effects

DETAILED DESCRIPTION:
Background: Plantar warts are a common dermatological condition caused by human papillomavirus infection. They can be painful and negatively impact quality of life. Many treatments exist but there is lack of consensus on the optimal approach.

Objectives:

Primary objective: To compare the efficacy of 980nm diode laser versus liquid nitrogen cryotherapy for clearing plantar warts, as measured by the complete clearance rate at 4 weeks post-treatment.

Secondary objectives: To evaluate and compare pain levels during treatment procedures and adverse events between both groups.

Study design: Randomized, double-blind clinical trial.

Participants: 32 patients aged 18-65 years old with 1-3 plantar warts located on weight-bearing areas of the foot.

Interventions:

Laser group: 980nm diode laser applied to each wart for 5 seconds at 2W power and 1mm spot size. 4 sessions at weekly intervals.

Cryotherapy group: Liquid nitrogen sprayed on each wart using a standardised technique. Freeze-thaw cycle repeated up to 3 times per wart per session. 4 sessions at weekly intervals.

Main outcomes:

Complete clearance rate of plantar warts at 4 weeks treatment session. Assessed by physical examination.

Pain during procedure measured with Visual Analogue Scale (VAS). Adverse events monitored during follow-up.

Randomization and blinding: Subjects will be randomly allocated to each group with a 1:1 ratio. Investigators assessing outcomes will be blinded to group assignment.

Analysis: Intention-to-treat analysis will be performed. Chi-squared test will compare clearance rates. T-test will compare pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recalcitrant, mosaic and simple HPV

Exclusion Criteria:

* Diabetic, ischaemic and immunosuppressed patients
* Patients with cold intolerance
* Patients with any of the following conditions (blood dyscrasias of unknown origin, cryoglobulinaemia, cryofibrinogenemia, collagen or autoimmune disease)
* Patients who do not sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Skin pattern | 7 days from first application
  Interrupted plantar lines with irregularly distributed dots.classifies the severity in 3 degrees, from the absence of alterations (0) to the extensive presence of interrupted lines and irregular spots in the plantar skin pattern (3).

SECONDARY OUTCOMES:
VAS scale | 7 days from first application
  It is a tool to allow the patient to evaluate the intensity of the pain on a visual scale of 0-10, where 0 is nothing and 10 is unbearable, being a subjective evaluation.
complications | 7 days from first application
  complications including the possibility of recurrence, discomfort or pain during or after treatment, risk of infection at the treated site, potential for scarring or changes in skin appearance, hypersensitivity or allergies to the drugs used, changes in skin pigmentation, and in rare cases, possibility of damage to surrounding structures such as nerves or blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ferrer-Torregrosa, Dr., Study Director — FundaciónUcv
Locations (2):
- Studio di Podologia Dr.Secolo, Catania, Sicily, Italy
- Clinicas UCV, Valencia, València, Spain

REFERENCES:
- [Result] Liu JJ, Li HT, Ren YY, Yang F, Cheng ZH, Xia TB, Liu JL, Cao XJ, Lu SC. Long-pulsed neodymium-doped yttrium-aluminum-garnet laser versus cryotherapy for the treatment of cutaneous warts: A randomized controlled trial. J Am Acad Dermatol. 2022 Dec;87(6):1328-1335. doi: 10.1016/j.jaad.2020.09.085. Epub 2020 Oct 5. PMID 33031838